CLINICAL TRIAL: NCT00021463
Title: Phase II, Randomized, Open-Label Study of Switching to Protease Inhibitor-Sparing Regimens for Improvement of Metabolic Abnormalities
Brief Title: Changing to Nonprotease Inhibitor Treatment to Improve Side Effects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Purpose: Treatment
Other Study IDs: ACTG A5103; AACTG A5103
Record Dates: First submitted 2001-07-14; First posted 2001-08-31 (Estimated); Last update posted 2011-02-28 (Estimated); Status verified 2003-01

CONDITIONS: HIV Infections; Lipodystrophy
Keywords: Nevirapine; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Triglycerides; abacavir; efavirenz; Lipoproteins, LDL Cholesterol
MeSH Terms: conditions — HIV Infections; Lipodystrophy | interventions — abacavir; Lamivudine; Zidovudine; efavirenz; Nevirapine

INTERVENTIONS:
Drug: Abacavir sulfate, Lamivudine and Zidovudine
Drug: Abacavir sulfate
Drug: Efavirenz
Drug: Nevirapine

SUMMARY:
The purpose of this study is to learn whether changing from a type of anti-HIV drug called a protease inhibitor (PI) to another type of anti-HIV drug will help to lower the amount of fats or sugars in the blood.

PIs have been effective at keeping HIV viral load (amount of HIV in the blood) down. However, some people who take PIs have higher than normal levels of fats and/or sugars in the blood. Doctors believe that switching to anti-HIV drugs that do not contain PIs will improve the abnormal side effects. This study will test 3 different combinations of non-PI drugs to see which may improve side effects while keeping viral loads low.

DETAILED DESCRIPTION:
Protease inhibitor (PI)-containing antiretroviral regimens are potent suppressors of HIV replication. Increasingly, metabolic abnormalities such as hypercholesterolemia and triglyceridemia are associated with PI use, reasons cited for switching to PI-sparing regimens. Yet optimal switch regimens that take into account both improvements in side effects and continued virologic suppression have not been defined. This study will compare the effect on chemical metabolic abnormalities of switching to an all nucleoside regimen versus dual nucleoside plus nonnucleoside reverse transcriptase inhibitor (NNRTI) therapy. Determining the effects of each regimen on chemical metabolic abnormalities and maintenance of virologic suppression will define which of the switch strategies being studied improves metabolic abnormalities without compromising viral suppression.

Patients are stratified on the basis of fasting non-HDL cholesterol and triglyceride levels and on ritonavir- or nonritonavir-containing pre-entry PI regimens. Patients are assigned randomly to add to their pre-entry regimen 1 of the following 3 treatments: Arm A - ABC; Arm B - NVP; or Arm C - EFV.

Patients discontinue pre-entry PIs after Day 14. Patients are followed to determine the effect of the maintenance regimens on fasting non-high-density lipoprotein (HDL), cholesterol, and triglycerides at Week 24. Fasting total cholesterol, HDL cholesterol, direct low-density lipoprotein, and triglycerides are measured at Weeks 12, 24, and 48. Fasting glucose, insulin, C-peptide, apolipoproteins A-1 and B, lipoprotein a, and homocysteine are measured at Weeks 24 and 48. Anthropometrics, body mass index, and body image are measured at Weeks 12, 24, and 48. HIV viral load is measured at Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, and 48. If HIV RNA stays below 200 copies/ml, therapy continues unchanged. If confirmed HIV RNA of 200 copies/ml or higher is found, an HIV genotype is obtained providing the viral load is sufficient to yield results, the best medical therapy is instituted (not supplied by the study), and off treatment/on study follow-up is continued. If patients are intolerant to a study drug, an alternate study drug (ABC, EFV, or NVP supplied by the study) is permitted and switched treatment/on study follow-up continued, or the best medical therapy is instituted (not supplied by the study), and off treatment/on study follow-up is continued. Patients are followed until the last patient enrolled has completed 48 weeks on study.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV infected.
* Are on their first combination of stable anti-HIV drugs (have not changed drugs for at least 6 months, except for reasons other than failing treatment or short interruptions of less than 7 days).
* Have 2 measurements of viral load (amount of HIV in the blood) during the 6 months before entering the study that are below 400 copies/ml by RT-PCR test or below 500 copies/ml by branched DNA test, measured at least 8 weeks apart.
* Have a viral load below 50 copies/ml within 30 days prior to entry.
* Have a CD4 cell count of 200 copies/ml or higher within 60 days of study entry.
* Are receiving medications and/or medications at certain doses that might interfere with the study.
* Are at least 13 years old and have signed consent of parent or guardian if under 18 years of age.
* Have a negative pregnancy test within 14 days of study entry, if a woman able to have children.
* Agree to use a barrier method of birth control, men and women, while receiving study drugs and for 3 months afterwards.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Are receiving high doses of testosterone. Low doses are allowed if received for 60 or more days before entering the study with no plans to change the dose during the first 24 weeks of the study.
* Have had treatment with any nonnucleoside reverse transcriptase inhibitor (NNRTI).
* Have had treatment with ABC.
* Are allergic to study drugs or any ingredient in them.
* Are pregnant or breast-feeding.
* Have used any HIV vaccine or drugs affecting the immune system within 30 days prior to entering the study.
* Have had systemic treatment for cancer within 30 days of entering the study.
* Have had systemic treatment with certain other drugs that may interfere with the study within 14 days of entering the study.
* Have a serious illness that required systemic treatment or a hospital stay unless treatment was completed at least 14 days prior to entering the study, or are on stable treatment, in the doctor's opinion, for at least 14 days prior to entering the study.
* Abuse drugs or alcohol.
* Have or suspect they have acute hepatitis within 30 days of entering the study.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 342
Dates: Primary Completion 2002-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wohl, Study Chair
Locations (11):
- United States (11):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Emory Univ, Atlanta, Georgia
  - Northwestern Univ Med School, Chicago, Illinois
  - The CORE Ctr, Chicago, Illinois
  - Boston Med Ctr, Boston, Massachusetts
  - Brigham and Women's Hosp, Boston, Massachusetts
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Univ of Pennsylvania, Philadelphia, Pennsylvania
  - Univ of Pittsburgh, Pittsburgh, Pennsylvania